CLINICAL TRIAL: NCT01178814
Title: A Prospective Trial of Revlimid® in Transfusion Dependent Patients With Non-del (5q) Low/Intermediate-1 Risk Myelodysplastic Syndrome
Brief Title: Revlimid in Transfusion Dependent Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAF2696
Record Dates: First submitted 2010-08-06; First posted 2010-08-10 (Estimated); Results first posted 2021-07-20 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Revlimid (Experimental): Revlimid (Lenalidomide) capsule taken orally once a day
  Interventions: Drug: Revlimid (Lenalidomide)

INTERVENTIONS:
Drug: Revlimid (Lenalidomide) — The starting dose will be 10 mg days 1-28 with the first dose reduction going to 5 mg days 1-28 of a 28 day cycle. Therapy will cease if there is no response after 12 weeks.
  Other Names: Revlimid

SUMMARY:
This is a prospective trial of Revlimid for subjects who have a blood cell cancer called myelodysplastic syndrome (MDS). Cells in their marrow make proteins through messages that are carried from the genes. The amount of the message tells researchers if the protein it is going to make is high or low. This is known as expression of genes. The purpose of this study is to conduct a prospective trial testing the idea that expression of specific genes can help to predict which patients will respond to study drug administration with Revlimid (lenalidomide).

DETAILED DESCRIPTION:
The first Revlimid® study reported by List et al included all transfusion dependent MDS patients, but given the early experience which showed a better response in del(5q) patients and those with lower risk disease, more patients belonging to this category were entered on the trial. The subsequent multi-center studies were focused entirely on the low/Int-1 patients who were transfusion dependent. In the present study, we would like to recapitulate the initial study by only treating the transfusion dependent, low and intermediate-1 risk MDS patients without deletion (5q). Since the predictive assay is most applicable for the non-del(5q) patients, and to avoid confusion resulting from an admixture of patients with del(5q) for whom the drug is already FDA approved, we have elected to restrict this clinical trial to only the non-del(5q) patients.

In the present study, only the non-del(5q) transfusion dependent, low and intermediate-1 risk MDS patients will be treated with single agent Revlimid®. All patients will have their pre-therapy bone marrows studied by gene expression microarray, Luminex bead assay, and real-time PCR.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Age ≥ 21 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* A confirmed diagnosis (using standard FAB criteria) of a myelodysplastic syndrome with low/Int-1 risk and with a non-del(5q) karyotype must be established.
* Patients must have transfusion dependence (at least 2 units within 8 weeks prior to starting therapy).
* All transfusion dependent non-del(5q) low/Int-1 risk patients will be eligible for treatment with Revlimid®
* Newly diagnosed as well as previously treated patients will be eligible
* Patients with primary de novo or secondary MDS will be eligible
* All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study.
* ECOG performance status of 0-2 at study entry (see Appendix II).
* Laboratory test results within these ranges:

  * Absolute neutrophil count > 250/uL
  * Platelet count > 30,000/uL
  * Serum creatinine ≤ 2.0 mg/dL
  * Total bilirubin ≤ 1.5 mg/dL
  * AST (SGOT) and ALT (SGPT) ≤ 3 x ULN
  * BUN ≤ 2 x ULN
* Disease free of prior malignancies for ≥ 2 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Any clinically significant cardiac disease, including congestive heart failure
* Liver function studies including SGOT/SGPT > 3 x ULN
* Clinically significant renal disease.
* Any previous chemotherapy, hematopoietic growth factors, erythropoietin, or cytokines within 4 weeks of starting treatment. Note: prior therapy with G-CSF within 4 weeks is allowed.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to thalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Any prior use of lenalidomide. (Patients with prior therapy with thalidomide will be eligible as long as at least 4 weeks have elapsed between end of the drug and accrual on the present trial)
* Concurrent use of other anti-cancer agents or treatments.
* Known positive for HIV or infectious hepatitis, type B or C.
* Life expectancy < 3 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Heaney, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Revlimid
Started | 57
Completed | 57
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Revlimid
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 37
  More than one race | 0
  Unknown or Not Reported | 17
Region of Enrollment [Number; unit: participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Response Signature in Transfusion Dependent MDS Patients
Description: The trial will be testing the Revlimid® (lenalidomide) response signature in patients who have transfusion dependent, non-del(5q), low and intermediate-1 risk myelodysplastic syndromes (MDS) in order to confirm the predictive value of the signature and to establish the boundaries of the z-score which can be used to pre-select patients in future clinical studies. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Up to 12 weeks from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Revlimid
Number analyzed (Participants) | 57
Participants
  No response | 24
  Delayed response | 1
  Complete Response (CR) | 17
  Partial Response (PR) | 6
  Other response | 9

ADVERSE EVENTS:
Time Frame: Up to 3 months
Arm/Group | Revlimid
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 3/57
Other Adverse Events (participants affected / at risk) | 8/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Revlimid (N=57)
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Revlimid (N=57)
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Diarrhea (Gastrointestinal disorders) | 4
Platelet count abnormality (Investigations) | 4
Rash (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-10-29): https://cdn.clinicaltrials.gov/large-docs/14/NCT01178814/Prot_SAP_000.pdf